CLINICAL TRIAL: NCT04454554
Title: Prevalence of Pulmonary Embolism (PE) Among Patients Referred to Emergency Departments for Dyspnea on Exertion
Brief Title: Prevalence of Pulmonary Embolism in Patients With Dyspnea on Exertion (PEDIS)
Acronym: PEDIS
Status: Completed | Type: Observational
Sponsor: Arianna Anticoagulazione Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: FAA O4 5-2018 (PEDIS)
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Pulmonary Embolism
Keywords: Dyspnea; Pulmonary embolism
MeSH Terms: conditions — Pulmonary Embolism; Dyspnea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PEDIS Study is an observational, cross-sectional, multicenter Italian study conducted in a consecutive series of patients who refer to the Emergency Departments (either spontaneously or sent by their attending physicians) for the recent (less than one months) development of exertional dyspnea.

The general aim of the study is to assess the prevalence of PE in the overall population referring to the Emergency Departments without potential explanations for dyspnea

DETAILED DESCRIPTION:
PEDIS Study is an observational, cross-sectional, multicenter and no Profit Study.

600 consecutive patients referring to the Emergency Departments of the participating centers because they have developed one or more episodes of exertional dyspnea since less than one month will be enrolled. All eligible patients will be interviewed and examined by trained study physicians. The presence of already known potential explanations for the dyspnea will be assessed. In addition, symptoms of the lower extremities will be elicited, as well as the presence of risk factors for venous thromboembolism (VTE).

The presence or absence of pulmonary embolism will be assessed with the use of a validated algorithm based on pre-test clinical probability and D-dimer result. In patients in whom the pre-test clinical probability is low and the D-dimer result is negative, no further testing will be done, and PE will be considered excluded. In patients with high clinical probability, positive D-dimer result, or both, computed tomography (CT) pulmonary angiography will be performed

The primary study objective is to evaluate Prevalence of PE in the overall population

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 and younger than 75
* Recent (less than one month) development of exertional dyspnea
* Able to provide informed consent

Exclusion Criteria:

* Anticoagulation required for other indications
* Contraindication to CT angiography (allergy to the contrast dye, severe renal failure [creatinine clearance < 30 ml/min])
* Involvement in simultaneous clinical trials
* Unable to provide their written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who refer to the Emergency Departments of the participating centers will be eligible for the study provided they are older than 18 and younger than 75 years, and have developed one or more episodes of exertional dyspnea since less than one month.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of PE in the overall population | From the first day of enrollment up to 104 weeks
  Prevalence of Pulmonary Embolism in patient with high pre-test clinical probability and/or positive D-dimer without potential explanations for the dyspnea who underwent computed tomography pulmonary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Bova, MD, Study Director — Azienda Ospedaliera di Cosenza
Locations (1):
- Azienda Ospedalier di Cosenza "SS.Annunziata", Cosenza, Italy

REFERENCES:
- [Derived] Prandoni P, Lensing AWA, Prins MH, Ciammaichella M, Pirillo S, Pace F, Zalunardo B, Bottino F, Ageno W, Muiesan ML, Forlin M, Depietri L, Bova C, Costantini N, Caviglioli C, Migliaccio L, Noventa F, Levi M, Davidson BL, Palareti G; Pulmonary Embolism Dyspnea Italian Study (PEDIS) Investigators. Prevalence of pulmonary embolism among patients with recent onset of dyspnea on exertion. A cross-sectional study. J Thromb Haemost. 2023 Jan;21(1):68-75. doi: 10.1016/j.jtha.2022.09.007. Epub 2022 Dec 22. PMID 36695397

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT04454554/Prot_SAP_000.pdf